CLINICAL TRIAL: NCT02407418
Title: The Effects of Lumbosacral Manipulation on Isokinetic Strength of the Knee Extensors and Flexors
Brief Title: The Effects of Spinal Manipulation on Thigh Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grant Sanders (Other)
Responsible Party: Sponsor-Investigator, Grant Sanders, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-0280-F1V
Record Dates: First submitted 2015-03-23; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Subluxation of Joint of Lumbar Spine
Keywords: spinal manipulation; muscle strength dynamometer; muscle strength
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal Manipulation (Active Comparator): In a repeated measures, crossover design, all subjects received spinal manipulation during the second or third session. The selection of spinal manipulation or sham was randomized.
  Interventions: Other: Spinal Manipulation
- Sham Manipulation (Sham Comparator): In a repeated measures, crossover design, all subjects received the sham manipulation during the second or third session. The selection of spinal manipulation or sham was randomized.
  Interventions: Other: Sham Manipulation

INTERVENTIONS:
Other: Spinal Manipulation — Side-posture, high-velocity low-amplitude spinal manipulation targeting the lumbar spine and sacroiliac joints
  Arms: Spinal Manipulation
Other: Sham Manipulation — A simulated lumbar spine manipulation in which no vertebral contact was made
  Arms: Sham Manipulation

SUMMARY:
The purpose of this study was to investigate the effects of chiropractic low back adjustments on thigh muscle strength. Force production was measured during different types of muscle contractions with a device called an isokinetic dynamometer. The study included 21 college-aged subjects who did not have any pain and had never received chiropractic treatment with spinal manipulation. During two separate sessions, subjects' thigh muscle forces were recorded while performing maximal muscle contractions on the isokinetic dynamometer. Baseline measurements of muscle force were acquired before either treatment form of spinal manipulation or a sham spinal manipulation, followed by identical muscle force measurements within five and twenty minutes post-treatment.

DETAILED DESCRIPTION:
Spinal manipulation is a therapeutic procedure employed by various healthcare practitioners for alleviating acute and chronic musculoskeletal complaints. This form of treatment is also delivered to enhance the performance and augment the rehabilitation of athletes. However, despite research findings alleging the strength-modulating effects of spinal manipulation alongside numerous professional athletes' positive anecdotal claims concerning its results, the physiological processes to explain its effects remain largely unexplained. Therefore, the purpose of this work was to investigate the effects of spinal manipulation in a college-aged sample population.

This study examined the effect of spinal manipulation delivered to the lumbosacral region on concentric force production of the knee extensors and flexors. A randomized, controlled, single-blind repeated measures design was utilized with 21 subjects. Isometric and isokinetic peak torques (Nm) were recorded during two separate session while subjects performed maximal voluntary contractions post-treatment of either spinal manipulation or a sham manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20 to 35 years
* Asymptomatic with regard to low back, pelvic or lower extremity pain

Exclusion Criteria:

* Previously received spinal manipulation from a chiropractor or other health care provider
* Contraindications to lumbar spine manipulation (such as fractures, lumbar disc herniation, abdominal aortic aneurysm or cauda equina syndrome)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in isometric and isokinetic peak torques compared to baseline | Baseline peak torque measurements were acquired before either treatment form of lumbosacral manipulation or sham manipulation, followed by identical peak torque measurements recorded within 5 minutes and at 20 minutes post-treatment
  Peak torque measurements were recorded in newton meters (Nm) while subjects performed maximal voluntary contractions of concentric knee extension and flexion during a randomized protocol of isometric and isokinetic contractions, all of which measured with an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Grant D Sanders, D.C., Principal Investigator — University of Kentucky

REFERENCES:
- [Background] Hurwitz EL. Epidemiology: spinal manipulation utilization. J Electromyogr Kinesiol. 2012 Oct;22(5):648-54. doi: 10.1016/j.jelekin.2012.01.006. Epub 2012 Jan 29. PMID 22289432
- [Background] Pickar JG. Neurophysiological effects of spinal manipulation. Spine J. 2002 Sep-Oct;2(5):357-71. doi: 10.1016/s1529-9430(02)00400-x. PMID 14589467
- [Background] Miners AL. Chiropractic treatment and the enhancement of sport performance: a narrative literature review. J Can Chiropr Assoc. 2010 Dec;54(4):210-21. PMID 21120012
- [Background] Grindstaff TL, Hertel J, Beazell JR, Magrum EM, Ingersoll CD. Effects of lumbopelvic joint manipulation on quadriceps activation and strength in healthy individuals. Man Ther. 2009 Aug;14(4):415-20. doi: 10.1016/j.math.2008.06.005. Epub 2008 Sep 20. PMID 18805726
- [Background] Hillermann B, Gomes AN, Korporaal C, Jackson D. A pilot study comparing the effects of spinal manipulative therapy with those of extra-spinal manipulative therapy on quadriceps muscle strength. J Manipulative Physiol Ther. 2006 Feb;29(2):145-9. doi: 10.1016/j.jmpt.2005.12.003. PMID 16461174
- [Background] Suter E, McMorland G, Herzog W, Bray R. Conservative lower back treatment reduces inhibition in knee-extensor muscles: a randomized controlled trial. J Manipulative Physiol Ther. 2000 Feb;23(2):76-80. PMID 10714531
- [Background] Suter E, McMorland G, Herzog W, Bray R. Decrease in quadriceps inhibition after sacroiliac joint manipulation in patients with anterior knee pain. J Manipulative Physiol Ther. 1999 Mar-Apr;22(3):149-53. doi: 10.1016/S0161-4754(99)70128-4. PMID 10220713
- [Background] Botelho MB, Andrade BB. Effect of cervical spine manipulative therapy on judo athletes' grip strength. J Manipulative Physiol Ther. 2012 Jan;35(1):38-44. doi: 10.1016/j.jmpt.2011.09.005. Epub 2011 Nov 10. PMID 22079053
- [Background] Fernandez-Carnero J, Fernandez-de-las-Penas C, Cleland JA. Immediate hypoalgesic and motor effects after a single cervical spine manipulation in subjects with lateral epicondylalgia. J Manipulative Physiol Ther. 2008 Nov-Dec;31(9):675-81. doi: 10.1016/j.jmpt.2008.10.005. PMID 19028251
- [Background] Paungmali A, Vicenzino B, Smith M. Hypoalgesia induced by elbow manipulation in lateral epicondylalgia does not exhibit tolerance. J Pain. 2003 Oct;4(8):448-54. doi: 10.1067/s1526-5900(03)00731-4. PMID 14622665
- [Background] Abbott JH, Patla CE, Jensen RH. The initial effects of an elbow mobilization with movement technique on grip strength in subjects with lateral epicondylalgia. Man Ther. 2001 Aug;6(3):163-9. doi: 10.1054/math.2001.0408. PMID 11527456
- [Background] Giggey K, Tepe R. A pilot study to determine the effects of a supine sacroiliac orthopedic blocking procedure on cervical spine extensor isometric strength. J Chiropr Med. 2009 Jun;8(2):56-61. doi: 10.1016/j.jcm.2008.11.002. PMID 19646387
- [Background] Keller TS, Colloca CJ. Mechanical force spinal manipulation increases trunk muscle strength assessed by electromyography: a comparative clinical trial. J Manipulative Physiol Ther. 2000 Nov-Dec;23(9):585-95. doi: 10.1067/mmt.2000.110947. PMID 11145798
- [Background] Suter E, McMorland G. Decrease in elbow flexor inhibition after cervical spine manipulation in patients with chronic neck pain. Clin Biomech (Bristol). 2002 Aug;17(7):541-4. doi: 10.1016/s0268-0033(02)00025-6. PMID 12206946
- [Background] Wang SS, Meadows J. Immediate and carryover changes of C5-6 joint mobilization on shoulder external rotator muscle strength. J Manipulative Physiol Ther. 2010 Feb;33(2):102-8. doi: 10.1016/j.jmpt.2009.12.006. PMID 20170775
- [Background] Panton LB, Figueroa A, Kingsley JD, Hornbuckle L, Wilson J, St John N, Abood D, Mathis R, VanTassel J, McMillan V. Effects of resistance training and chiropractic treatment in women with fibromyalgia. J Altern Complement Med. 2009 Mar;15(3):321-8. doi: 10.1089/acm.2008.0132. PMID 19249999
- [Background] Morningstar MW. Strength gains through lumbar lordosis restoration. J Chiropr Med. 2003 Autumn;2(4):137-41. doi: 10.1016/S0899-3467(07)60077-9. PMID 19674610
- [Background] de Almeida BS, Sabatino JH, Giraldo PC. Effects of high-velocity, low-amplitude spinal manipulation on strength and the basal tonus of female pelvic floor muscles. J Manipulative Physiol Ther. 2010 Feb;33(2):109-16. doi: 10.1016/j.jmpt.2009.12.007. PMID 20170776
- [Background] Chilibeck PD, Cornish SM, Schulte A, Jantz N, Magnus CR, Schwanbeck S, Juurlink BH. The effect of spinal manipulation on imbalances in leg strength. J Can Chiropr Assoc. 2011 Sep;55(3):183-92. PMID 21886280
- [Background] Knapik JJ, Wright JE, Mawdsley RH, Braun J. Isometric, isotonic, and isokinetic torque variations in four muscle groups through a range of joint motion. Phys Ther. 1983 Jun;63(6):938-47. doi: 10.1093/ptj/63.6.938. PMID 6856681
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Sole G, Hamren J, Milosavljevic S, Nicholson H, Sullivan SJ. Test-retest reliability of isokinetic knee extension and flexion. Arch Phys Med Rehabil. 2007 May;88(5):626-31. doi: 10.1016/j.apmr.2007.02.006. PMID 17466732
- [Background] Drouin JM, Valovich-mcLeod TC, Shultz SJ, Gansneder BM, Perrin DH. Reliability and validity of the Biodex system 3 pro isokinetic dynamometer velocity, torque and position measurements. Eur J Appl Physiol. 2004 Jan;91(1):22-9. doi: 10.1007/s00421-003-0933-0. Epub 2003 Sep 24. PMID 14508689
- [Background] Todd G, Gorman RB, Gandevia SC. Measurement and reproducibility of strength and voluntary activation of lower-limb muscles. Muscle Nerve. 2004 Jun;29(6):834-42. doi: 10.1002/mus.20027. PMID 15170616
- [Background] Akebi T, Saeki S, Hieda H, Goto H. Factors affecting the variability of the torque curves at isokinetic trunk strength testing. Arch Phys Med Rehabil. 1998 Jan;79(1):33-5. doi: 10.1016/s0003-9993(98)90204-0. PMID 9440414
- [Background] Frost LR, Gerling ME, Markic JL, Brown SH. Exploring the effect of repeated-day familiarization on the ability to generate reliable maximum voluntary muscle activation. J Electromyogr Kinesiol. 2012 Dec;22(6):886-92. doi: 10.1016/j.jelekin.2012.05.005. Epub 2012 Jun 20. PMID 22726611
- [Background] Pickar JG, Bolton PS. Spinal manipulative therapy and somatosensory activation. J Electromyogr Kinesiol. 2012 Oct;22(5):785-94. doi: 10.1016/j.jelekin.2012.01.015. Epub 2012 Feb 19. PMID 22349622
- [Background] Haavik H, Murphy B. The role of spinal manipulation in addressing disordered sensorimotor integration and altered motor control. J Electromyogr Kinesiol. 2012 Oct;22(5):768-76. doi: 10.1016/j.jelekin.2012.02.012. Epub 2012 Apr 6. PMID 22483612
- [Background] Korr IM. Somatic dysfunction, osteopathic manipulative treatment, and the nervous system: a few facts, some theories, many questions. J Am Osteopath Assoc. 1986 Feb;86(2):109-14. No abstract available. PMID 3753964
- [Background] Dishman JD, Bulbulian R. Spinal reflex attenuation associated with spinal manipulation. Spine (Phila Pa 1976). 2000 Oct 1;25(19):2519-24;discussion 2525. doi: 10.1097/00007632-200010010-00015. PMID 11013505
- [Background] Budgell BS. Reflex effects of subluxation: the autonomic nervous system. J Manipulative Physiol Ther. 2000 Feb;23(2):104-6. doi: 10.1016/s0161-4754(00)90076-9. PMID 10714536
- [Background] Bolton PS. Reflex effects of vertebral subluxations: the peripheral nervous system. An update. J Manipulative Physiol Ther. 2000 Feb;23(2):101-3. doi: 10.1016/s0161-4754(00)90075-7. PMID 10714535
- [Background] Taylor HH, Murphy B. Altered sensorimotor integration with cervical spine manipulation. J Manipulative Physiol Ther. 2008 Feb;31(2):115-26. doi: 10.1016/j.jmpt.2007.12.011. PMID 18328937
- [Background] DeVocht JW, Pickar JG, Wilder DG. Spinal manipulation alters electromyographic activity of paraspinal muscles: a descriptive study. J Manipulative Physiol Ther. 2005 Sep;28(7):465-71. doi: 10.1016/j.jmpt.2005.07.002. PMID 16182019
- [Background] Colloca CJ, Keller TS. Electromyographic reflex responses to mechanical force, manually assisted spinal manipulative therapy. Spine (Phila Pa 1976). 2001 May 15;26(10):1117-24. doi: 10.1097/00007632-200105150-00005. PMID 11413422
- [Background] Haavik-Taylor H, Murphy B. Cervical spine manipulation alters sensorimotor integration: a somatosensory evoked potential study. Clin Neurophysiol. 2007 Feb;118(2):391-402. doi: 10.1016/j.clinph.2006.09.014. Epub 2006 Nov 29. PMID 17137836
- [Background] Lehman G. Kinesiological research: the use of surface electromyography for assessing the effects of spinal manipulation. J Electromyogr Kinesiol. 2012 Oct;22(5):692-6. doi: 10.1016/j.jelekin.2012.02.010. Epub 2012 Mar 15. PMID 22425147
- [Background] Colloca CJ, Keller TS, Gunzburg R. Neuromechanical characterization of in vivo lumbar spinal manipulation. Part II. Neurophysiological response. J Manipulative Physiol Ther. 2003 Nov-Dec;26(9):579-91. doi: 10.1016/j.jmpt.2003.08.004. PMID 14673407
- [Background] Colloca CJ, Keller TS, Gunzburg R, Vandeputte K, Fuhr AW. Neurophysiologic response to intraoperative lumbosacral spinal manipulation. J Manipulative Physiol Ther. 2000 Sep;23(7):447-57. doi: 10.1067/mmt.2000.108822. PMID 11004648
- [Background] Krishnan C, Williams GN. Error associated with antagonist muscle activity in isometric knee strength testing. Eur J Appl Physiol. 2010 Jun;109(3):527-36. doi: 10.1007/s00421-010-1391-0. Epub 2010 Feb 20. PMID 20174928
- [Background] Krishnan C, Williams GN. Variability in antagonist muscle activity and peak torque during isometric knee strength testing. Iowa Orthop J. 2009;29:149-58. PMID 19742105